CLINICAL TRIAL: NCT01524718
Title: Internal Fixation of Hip Fractures Using Intraoperative Simultaneous Two Axis View
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MMC-twoaxis-001.il
Record Dates: First submitted 2012-01-10; First posted 2012-02-02 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Fracture Neck of Femur
Keywords: radiation; time surgery
MeSH Terms: conditions — Femoral Neck Fractures | interventions — X-Rays

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imaging with two X-ray image intensifiers (Experimental): There is no change in the procedure except for the imaging technique, while in the first group the X- ray image intensifier serves in the two planes, and being moved from one plane to the other, and in the second group the two devices are static in the same position, one in the AP plane and the other as the axial plane.
  Interventions: Radiation: Imaging with two X-ray image intensifiers
- Imaging with one X-ray image intensifier. (No Intervention): The X- ray image intensifier serves in the two planes, and being moved from one plane to the other

INTERVENTIONS:
Radiation: Imaging with two X-ray image intensifiers — Two fluoroscopy apparatus one in the AP plane and the other as the axial plane.
  Arms: Imaging with two X-ray image intensifiers

SUMMARY:
Hip fractures are one of the most frequent operated fractures procedures in orthopedics, with a world wide annual incidence of approximately 1.7 million. These fractures are associated with substantial morbidity and mortality. As populations age and life expectancy increases worldwide, the incidence of these fractures is likely to raise, expected to triple in the next 50 years. The use of fluoroscopy and resultant exposure to radiation, is an integral part of surgical procedures aiming to reduce and fixate the fractured femur. The risk of contracting cancer is significantly higher for an orthopedic surgeon as Hip surgery is a major slice of the total radiation dose. Optimal positioning and control of the imaging intensifier device may result in significant reduction of radiation dose and time and in substantial shortening of the procedure.

The investigators hypothesis is that this technique would substantially shorten procedure time and reduce unnecessary radiation exposure for both the patient and the medical staff. Furthermore, by using this technique the investigators can eliminate the need for fluoroscopy technician during the surgery, as there is no need to alternate fluoroscopy views.

ELIGIBILITY:
Inclusion Criteria:

* patients with intertrochanteric femoral fracture who are going to be operated by closed reduction and internal fixation with an intramedullary nail.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-10 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Time of surgery | 5 hours - operation time
  time of operation

SECONDARY OUTCOMES:
X-ray time during surgery | 5 hours - operation time
  radiation time
Accuracy of nail position | 5 hours - operation time
Accuracy of reduction | 5 hours - operation time

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel